CLINICAL TRIAL: NCT03188627
Title: A Single-centered, Non-randomized, Concurrent Control Study on Autologous Bronchial Basal Cell Transplantation for Treatment of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Autologous Bronchial Basal Cell Transplantation for Treatment of COPD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regend Therapeutics (Industry)
Collaborators: Southwest Hospital, China (Other); Tongji University (Other)
Responsible Party: Principal Investigator, Xiaotian Dai, principal investigator, Regend Therapeutics
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170206
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchial basal cells (Experimental): Transplantation of autologous bronchial basal cells
  Interventions: Biological: Bronchial basal cells
- Control (No Intervention): Conventional treatment

INTERVENTIONS:
Biological: Bronchial basal cells — Transplantation of autologous bronchial basal cells
  Arms: Bronchial basal cells

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is usually characterized by long-term poor airflow, resulting in chronic pulmonary heart disease, chronic respiratory failure or even death. For COPD patients, pulmonary bronchus structures are damaged and cannot be repaired by recent clinical methods so far. This study intends to carry out a single-centered and non-randomized phase I/II clinical trial with concurrent controls to investigate whether bronchial basal cells can regenerate damaged lung tissue. During the treatment, bronchial basal cells will be isolated from patients' own bronchi and expanded in vitro. After careful characterization, expanded cells will be transplanted autologously into the lesion by fiberoptic bronchoscopy. The safety and efficacy of the treatment will be monitored by measuring the key clinical indicators.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 to 75;
* Diagnosed with COPD according the guideline (a. with symptoms of productive cough, sputum production or shortness of breath; b. with poor airflow as indicated by FEV1<70% predicted value and FEV1/FVC < 0.7 in pulmonary function test; c. with exclusion of other pulmonary disease by CT or blood examination.);
* Current smoker or ex-smoker with a history of no less than 10 years or 10 packs/year;
* Tolerant to bronchofiberscope;
* Written informed consent signed.

Exclusion Criteria:

* Pregnant or lactating women;
* Patients positive for syphilis, HIV;
* Patients with malignant tumor;
* Patients with serious significant pulmonary infection and need anti-infection treatment;
* Patients with serious heart disease(NYHA class Ⅲ-Ⅳ);
* Patients with a history of abusing alcohol and illicit drug;
* Patients participated in other clinical trials in the past 3 months;
* Patients assessed as inappropriate to participate in this clinical trial by investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Indicators for safety | 1-6 months
  Measured by blood routine test, urine routine test and blood chemistry panels
Diffusion capacity of CO (DLCO) | 1-6 months
  One of the indicators in pulmonary function test, the extent to which oxygen passes from the air sacs of the lungs into the blood

SECONDARY OUTCOMES:
The ratio of forced expiratory volume in the first one second to the forced vital capacity (FEV1/FVC) | 1-6 months
  One of the indicators in pulmonary function test, representing the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration to the full vital capacity
Maximum mid-expiratory flow (MMF) | 1-6 months
  One of the indicators in pulmonary function test, standing for maximal (mid-)expiratory flow and is the peak of expiratory flow as taken from the flow-volume curve and measured in liters per second
Maximum voluntary ventilation (MVV) | 1-6 months
  One of the indicators in pulmonary function test, measuring the maximum amount of air that can be inhaled and exhaled within one minute
Forced expiratory volume in one second (FEV1) | 1-6 months
  One of the indicators in pulmonary function test, a marker to assess airway obstruction
6-minute-walk test (6MWT) | 1-6 months
  An indicator to evaluate the exercise function of patients with moderate or severe pulmonary heart diseases
Modified medical research council (MMRC) chronic dyspnea scale | 1-6 months
  An indicator to evaluate the level of dyspnea
St. George's respiratory questionnaire (SGRQ) scale | 1-6 months
  A questionnaire to assess life quality affected by the respiratory problems
Imaging of lung by high resolution computed tomography (HR-CT) | 1-6 months
  HR-CT images of lung will be analyzed to indicate the pulmonary structure.
Forced vital capacity (FVC) | 1-6 months
  One of the indicators in pulmonary function test, indicating the maximum amount of air a person can expel from the lungs after a maximum inhalation

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of the Third Military University, PLA (Southwest Hospital), Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zuo W, Zhang T, Wu DZ, Guan SP, Liew AA, Yamamoto Y, Wang X, Lim SJ, Vincent M, Lessard M, Crum CP, Xian W, McKeon F. p63(+)Krt5(+) distal airway stem cells are essential for lung regeneration. Nature. 2015 Jan 29;517(7536):616-20. doi: 10.1038/nature13903. Epub 2014 Nov 12. PMID 25383540